CLINICAL TRIAL: NCT00177710
Title: Pharmacokinetic Profile of Inhaled Liposomal Amphotericin B in Lung Transplant Recipients - Ambisome Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Shahid Husain, MD, UPMC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB# 0408180; NCT00235638 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Lung Transplantation; Fungal Infections
MeSH Terms: conditions — Mycoses | interventions — Amphotericin B

INTERVENTIONS:
Drug: Amphotericin B

SUMMARY:
The purpose of this study is to determine the steady state concentrations of inhaled liposomal amphotericin B (Ambisome®) in lung transplant recipients via aerosolized nebulization.

DETAILED DESCRIPTION:
Each subject will receive 1 mg/kg/day of inhaled Ambisome® for four days prior to the BAL (bronchoalveolar lavage) procedure. The dosage of 1 mg/kg was calculated by extrapolating the dosage of 1.6 mg/kg for the surface area of the rat lung to the human lung surface area in a 60 kg individual.

All four doses will be given in the presence of a physician and/or study coordinator. The forty eight subjects will be randomized such that six subjects undergo the BAL at 1, 12, 24, 48, 72, 96, 120, and 168 hours after the last dose of inhaled Liposomal amphotericin B (AmBisome®).

A blood sample (5 ml) will be obtained prior to the fourth dose of study medication and on the day of bronchoscopy (pseudo steady state trough). Concentrations of amphotericin in the serum, and bronchoalveolar lavage will be measured at pre-specified intervals after administration of liposomal amphotericin B (AmBisome®) in lung transplant recipients undergoing routine bronchoscopy as mentioned earlier.

A 5 ml blood sample will be recovered at the time of bronchoscopy for the purpose of determination of serum amphotericin B concentration and for the determination of serum urea concentration.

The bronchoscopy and bronchoalveolar lavage of subjects is done as a part of routine transplant care. Subjects will be followed for the follow-up of results of bronchoscopy at the interval deemed necessary by their transplant pulmonologist. The samples (blood and bronchoalveolar samples) will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location (ID lab at 8th floor Scaife Hall). The investigators on this study will keep the samples indefinitely. Samples may be given to investigators outside of UPMC or may be utilized in future studies about infectious diseases. If the samples are given to investigators not associated with this study, the samples will be provided without any identifiers. No genetic testing will be done on the samples obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male and female lung transplant recipients at University of Pittsburgh Medical Center ≥ 18 years of age will be eligible for the study.
* Single or double lung transplant recipients
* Willing to be available at the testing center for 4 consecutive days
* Able to comprehend and complete informed consent

Exclusion Criteria:

* Pregnant women or women capable of bearing children, who will not perform a urine pregnancy test
* Nursing mothers
* Subjects with hypersensitivity to amphotericin deoxycholate or liposomal amphotericin
* Subjects with a past history of bronchospasm associated with aerosol drug use
* Subjects with active bacterial or viral infection as defined by the current use of non-prophylactic antibiotic anti-viral medications
* Subjects with a forced expiratory volume in 1 second (FEV1) < 30% predicted or forced vital capacity (FVC) < 30% will not receive study medication.
* Subjects requiring supplemental oxygen
* Receipt of inhalational or intravenous (IV) amphotericin B within last 30 days
* Subjects with known fungal infection as per Mycoses Study Group (MSG) criteria on therapy with antifungal drugs or diagnosed on the day of bronchoscopy
* Serum creatinine > 1.9 mg/dl on the day of screening
* Liver enzymes ALT/AST/alkaline phosphatase greater than two times the normal limit
* Concurrent intravenous aminoglycoside use
* Subject with fever > 38.2°C
* Subjects on mechanical ventilation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-01; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetic profile of liposomal amphotericin B achieved in the serum and epithelial lining fluid of the lung with four doses of liposomal amphotericin B administered via aerosolized nebulization in lung transplant recipients

SECONDARY OUTCOMES:
The purpose of this study is to determine the steady state concentrations of inhaled liposomal amphotericin B (Ambisome®) in lung transplant recipients via aerosolized nebulization.

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Husain, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States